CLINICAL TRIAL: NCT00901966
Title: Sun Exposure and Melanoma in Agricultural Workers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909143; 09-C-N143
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Melanoma
Keywords: Melanoma; Sun Exposure History; Agricultural Health Study; Sun Exposure
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Agricultural workers and spouses: Melanoma risk factors among Ag workers and spouses who use pesticides.

SUMMARY:
This K07 Career Development Award application is designed to expand Dr. Dennis career development from cancer etiology to cancer prevention and control. The career development plan rests on mentoring directed by experts in cancer prevention research and protected time to foster my professional development as an independent cancer control researcher. A unique population, the Agricultural Health Study (AHS) cohort, will be used to examine sun exposure, sun protection behavior, and factors affecting these behaviors regarding the risk of melanoma in private pesticide applicators (farmers) and their spouses.

The research plan proposed to examine skin melanoma within this prospective cohort of private applicators (mostly farmers) and their spouses in Iowa and North Carolina (the AHS) in association with environmental factors. Specific aim 1 examined the risk of melanoma in the AHS cohort using various existing measures of sun exposure adjusted for skin sensitivity and sun protection. Subsequently (for aim 2) qualitative research methods were used to design appropriate measures of sun exposure, sun protection behavior, and factors affecting these behaviors in private applicators and their spouses within the AHS based on the cohort analyses.

Now Aim 3 will be completed by conducting a nested case-control study of melanoma within the AHS cohort to examine in more detail sun exposure histories and protective behavior. The questionnaire was designed based on findings from the cohort analyses (aim 1) and qualitative methods (aim 2). The risk of melanoma will be examined regarding: a) the complex relationship of cumulative (sun exposure during each decade of life) and intermittent sun exposure (sunburns and sunny vacations), b) factors affecting behavior including attitudes about sun exposure and prevention, and c) the use of tanning salons and sunless tanning creams, particularly in spouses (expected to be rare overall).

The final aim is to use the results from the cohort and nested case-control studies to design a behavioral intervention, along with short computer automated telephone interview (CATI) that can be used in the whole AHS cohort or other farming populations. Funding for such studies will be sought through the R01) mechanism as an independent cancer control researcher. The behavioral intervention will be based on those factors that are the strongest risk factors for melanoma, highly prevalent, and easily modifiable. The behavioral intervention will be designed based on knowledge and skill gained from the Career Development Plan goals.

DETAILED DESCRIPTION:
This K07 Career Development Award application is designed to expand Dr. Dennis career development from cancer etiology to cancer prevention and control. The career development plan rests on mentoring directed by experts in cancer prevention research and "protected time" to foster my professional development as an independent cancer control researcher. A unique population, the Agricultural Health Study (AHS) cohort, will be used to examine sun exposure, sun protection behavior, and factors affecting these behaviors regarding the risk of melanoma in private pesticide applicators (farmers) and their spouses. The research plan proposed to examine skin melanoma within this prospective cohort of private applicators (mostly farmers) and their spouses in Iowa and North Carolina (the AHS) in association with environmental factors. Specific aim 1 examined the risk of melanoma in the AHS cohort using various existing measures of sun exposure adjusted for skin sensitivity and sun protection. Subsequently (for aim 2), qualitative research methods were used to design appropriate measures of sun exposure, sun protection behavior, and factors affecting these behaviors in private applicators and their spouses within the AHS based on the cohort analyses. Now Aim 3 will be completed by conducting a nested case-control study of melanoma within the AHS cohort to examine in more detail sun exposure histories and protective behavior. The questionnaire was designed based on findings from the cohort analyses (aim 1) and qualitative methods (aim 2). The risk of melanoma will be examined regarding: a) the complex relationship of cumulative (sun exposure during each decade of life) and intermittent sun exposure (sunburns and sunny vacations), b) factors affecting behavior including attitudes about sun exposure and prevention, and c) the use of tanning salons and sunless tanning creams, particularly in spouses (expected to be rare overall). The final aim is to use the results from the cohort and nested case-control studies to design a behavioral intervention, along with a short computer automated telephone interview (CATI) that can be used in the whole AHS cohort or other farming populations. Funding for such studies will be sought through the R01 mechanism as an independent cancer control researcher. The behavioral intervention will be based on those factors that are the strongest risk factors for melanoma, highly prevalent, and easily modifiable. The behavioral intervention will be designed based on knowledge and skill gained from the Career Development Plan goals.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Registered Agricultural Health Study (AHS) participants in Iowa

EXCLUSION CRITERIA:

* prior cancer diagnosis other than melanoma
* surrogates will not be used if a case has died before they are interviewed
* participants under 18 will not be included.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Members of the the AHS cohort -- registered private pesticide applicators (mostly farmers) and their spouses -- in Iowa.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2009-05-12 (Actual); Primary Completion 2010-10-31 (Actual); Study Completion 2013-02-13 (Actual)

PRIMARY OUTCOMES:
Prevalence of melanoma | After enrollment
  Diagnosis of melanoma after enrollment into Agricultural Health Study

CONTACTS AND LOCATIONS:
Overall Officials: Laura Beane-Freeman, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States